CLINICAL TRIAL: NCT05636579
Title: Phase 1, Multiple Dose, Open-Label Study to Assess the Safety and Tolerability of EO2002 Intracameral Injections With or Without Topical Ripasudil in the Treatment of Corneal Edema
Brief Title: Study to Assess Safety and Tolerability of Multiple Doses of EO2002
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Collaborators: Emmecell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VSH-003
Record Dates: First submitted 2022-11-08; First posted 2022-12-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Corneal Edema; Corneal Endothelial Dystrophy; Endothelial Dysfunction; Fuchs Dystrophy; Fuchs' Endothelial Dystrophy; Bullous Keratopathy; Pseudophakic Bullous Keratopathy; Corneal Edema Pseudophakic
MeSH Terms: conditions — Corneal Edema; Corneal Dystrophy, Posterior Polymorphous, 1; Fuchs' Endothelial Dystrophy | interventions — K-115

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EO2002 with Ripasudil (Experimental): EO2002 + topical Ripasudil daily, then reinjection at week 6 + topical Ripasudil daily
  Interventions: Biological: EO2002; Drug: Ripasudil
- EO2002 without Ripasudil (Experimental): EO2002 injection at Day 0 and re-injection at Week 6
  Interventions: Biological: EO2002

INTERVENTIONS:
Biological: EO2002 — Intracameral injection of magnetic human corneal endothelial cells (EO2002)
Drug: Ripasudil — Daily use of Ripasudil drops
  Arms: EO2002 with Ripasudil

SUMMARY:
The goal of this clinical study is to assess the safety of multiple intracameral injections of EO2002 with and without topical Ripasudil.

ELIGIBILITY:
Inclusion Criteria:

All ocular criteria apply to the study eye unless otherwise noted.

1. Age ≥ 18 years.
2. Subject is phakic or pseudophakic with a posterior chamber intraocular lens (lens in the bag or sulcus).
3. Symptomatic corneal edema associated with endothelial dysfunction which may be secondary to Fuchs' corneal dystrophy or pseudophakic bullous keratopathy.

Key Exclusion Criteria:

All ocular criteria apply to the study eye unless otherwise noted.

1. Other corneal disease
2. Anterior chamber intraocular lens
3. Sutured or scleral-fixated intraocular lens.
4. Macular disease that in the investigator and/or sponsor's opinion would limit the ability of the subject to demonstrate improvement in BCVA.
5. History of refractive surgery.
6. History of Vitrectomy
7. Descemet membrane detachment.
8. History of uveitis or other ocular inflammatory disease.
9. History of incisional glaucoma surgery (e.g.,trabeculectomy, glaucoma drainage implant).
10. IOP >21 or <7 mm Hg
11. Prior incisional eye surgery within 3 months prior to study treatment or penetrating or endothelial keratoplasty.

11. History of ocular neoplasm. 12. ETDRS BCVA in the fellow eye is worse than 35 letters (Snellen equivalent of 20/200).

13. Female who is pregnant, nursing, or planning to become pregnant, or who is of childbearing potential and not using a reliable means of contraception during the study.

14. Subject is currently participating in or has participated within the last 3 months in any other clinical trial of an investigational drug by ocular or systemic administration.

15. Any concomitant medical or psychological condition that could interfere with study participation or is otherwise not suitable for entry into the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-12-09 (Estimated); Study Completion 2025-12-09 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability of multiple doses of EO2002 | 32 weeks
  Incidence of Treatment-Emergent Adverse Events

SECONDARY OUTCOMES:
Central Corneal Thickness | 32 weeks
  Changes in CCT compared to baseline
Best Corrected Visual Acuity | 32 weeks
  Changes in BCVA compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Sanchez Huerta, MD, Principal Investigator — Asociacion para Evitar la Ceguera
Locations (1):
- Asociacion para Evitar la Ceguera en Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No